CLINICAL TRIAL: NCT07136740
Title: BioTenCer: a Randomized, Wait-list Controlled Study to Assess the Safety and Efficacy of the Cerebri-biofeedback Device as Preventive Treatment in Adult Participants With Frequent and Chronic Tension Type Headache.
Brief Title: BioTenCer: Biofeedback as Preventive Treatment in Tension Type Headache
Acronym: BioTenCer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other); University Hospital, Akershus (Other); Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HelseNTHF; 24/07853 (Other: Norwegian Medikal Products Agency)
Record Dates: First submitted 2025-03-17; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Tension Type Headache
Keywords: biofeedback; tension type headache; therapist independent treatment
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment group is randomized to receive biofeedback treatment for 12 weeks. The intervention arm- treatment-group will be offered contribute with in an extension phase: an additional 12 weeks of eDiary recordings if they are willing.
  Interventions: Device: Cerebri-TTH biofeedback; Other: headache diary
- wait-list group (Placebo Comparator): The wait-list group does not receive any specific treatment for 12 weeks but serves as an important basis for comparison to evaluate the treatment effect. This group will keep daily headache diary for 12 weeks. placebo group will be offered Cerebri-TTH biofeedback in extension phase.
  Interventions: Other: headache diary

INTERVENTIONS:
Device: Cerebri-TTH biofeedback — Cerebri-TTH biofeedback device is a therapist-independent home-based smartphone treatment application (app). Cerebri-TTH is a medical device in risk class IIa, according to MDR, and includes two non-invasive wireless sensors and a smartphone application. Both sensors shall be in contact with the skin: one sensor is applied on the index finger and measures heart rate (HR), heart rate variability (HRV) and peripheral skin temperature. The second sensor is applied on the trapezius muscle using adhesive electrodes and measures muscle tension. The sensors transmit the measurements to the user's smartphone where the user is instructed to perform a biofeedback session. The sensors are to be used for 10 minutes per session per day. The user can choose to use the device more frequently if desired - up to 6 sessions per day.
  Arms: Treatment group
Other: headache diary — Participants randomized to the wait-list arm, are instructed to keep daily eDairy entries for 12 weeks.
  The wait list control group will be offered active treatment for 12 weeks after the initial 12-week wait-list period is completed in an extension phase.

SUMMARY:
The purpose of this study is to test a therapist-independent home-based smartphone app-based biofeedback treatment in adults with tension type headache. The aim of the study is to assess the safety and performance of the Cerebri-TTH biofeedback device as a preventive treatment in adults with frequent and chronic tension type headache.

The primary endpoint of the study is the change in the mean Area-Under-the-headache-Curve (AUC) from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the placebo group.

DETAILED DESCRIPTION:
This trial, BioTenCer, is a clinical study to test the efficacy and safety of the app-based biofeedback treatment, Cerebri-TTH, for tension type headache in adults. Bodily signals that are thought to be associated with TTH are measured by sensors during biofeedback. During the treatment, one sensor is placed on the skin above the upper trapezius muscle fibers to measure shoulder and neck muscle tension and one sensor is attached to the index finger to measure peripheral skin temperature and heart rate variability. By getting on-screen feedback on the phone, the user can learn techniques to reduce muscle tension, and increase finger temperature and heart rate variability. Reduced muscle tension, as well as an increase in finger temperature and heart rate variability is a sign of relaxation and a deactivation of the autonomous nervous system, which can lead to less intensity and fewer days of TTH. The aim of the study is to investigate the safety and efficacy of biofeedback treatment using Cerebri-TTH compared to wait-list controls. In this study, the investigators will randomize 300 adults with frequent and chronic TTH. All participants will complete a minimum of 4 weeks of daily headache diary entries in the Cerebri-TTH app. This will serve as the "baseline" measurements. Subsequently, the participants will be randomized to either the treatment group or the wait-list group. The treatment group will conduct daily biofeedback sessions (one session has a duration of 10 minutes) for 12 weeks. The wait-list group does not receive any specific treatment for 12 weeks but serves as an important basis for comparison to evaluate the treatment effect. The wait list control group will be offered active treatment for 12 weeks after the initial 12-week wait-list period is completed in an extension phase. Similarly, the intervention arm can contribute with an additional 12 weeks of eDiary recordings if they are willing. Participants in both groups (the treatment group and the wait-list control group) must complete daily registrations in the headache diary included in the app. The primary endpoint of the study is the change in the mean Area-Under-the-headache-Curve (AUC) from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the placebo group. AUC is calculated from a curve of the duration and intensity of headaches. Secondary key endpoints include the change in intensity of TTH, the change in duration of TTH, the change in mean number of days with TTH, the change in consumption of acute medication for TTH and the number, of participants with at least 30%, 50%, 75% and 100% reduction in mean Area-Under-the headache Curve (AUC). Preventive treatments for TTH, both drug and non-drug, have limited effects and potentially numerous side effects. If the biofeedback app proves to be effective, it may represent a useful and viable treatment option for TTH patients, that is readily available and unlikely to cause unwanted side effects.

Number of Participants: the investigators will randomize 300 adult patients with TTH, with 150 participants randomized to each arm.

The study consists of two arms. There is a run-in screening period of 4 weeks for both arms, and a treatment/waitlist period of 12 weeks. Subsequently, an extended treatment period of 12 weeks is offered to the waitlist control group. The participants in the treatment are arm are asked to contribute to an additional 12 weeks of daily eDairy registration explore the headache status and safety aspects after ended biofeedback training. The total duration of study participation for each participant is 16 weeks for the intervention arm and for the wait-list control arm which includes the screening/inclusion visit, a run-in period of 4 weeks without study intervention, a 12-week treatment/waitlist period with 3 planned telephone follow-ups before a final visit. An additional 12 weeks extension is offered participants, and in such cases the final visit is placed at the end of the extension phase. Subjects will complete daily app-based biofeedback sessions of 10 minutes per session for 12 weeks as the study intervention

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age inclusive or older, at the time of signing the informed consent.
* A diagnosis of TTH according to the criteria of the International Classification of Headache Disorders 3rd edition (ICHD-3)
* History of at least 6 days or more with TTH per 28-day period in the 3 months prior to screening (as recalled by the subject).
* Frequency of at least 6 days or more with TTH per 28-day period, confirmed by daily diary entries in the baseline period.
* At least three months of experience with smartphone and access to an iOS or Android phone at home.
* Capability of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Onset of TTH (and migraine, if present) before the age of 50 years.
* The onset of TTH should be present for at least 1 year prior to inclusion.

Exclusion Criteria:

* Subject does not master a Scandinavian language at a level sufficient to fully understand the written and verbal study information.
* Subject is unable to differentiate TTH from other concomitant headaches.
* A history of more than 1 migraine attack per month on average in the last year, as recalled by the patient.
* Frequency of more than 1 migraine attack per month during the baseline period, as confirmed by daily diary entries.
* Subjects diagnosed with trigeminal autonomic cephalalgias and cranial neuralgias.
* Subjects with secondary headache conditions with the exception of medication overuse headache (MOH) as defined in the ICHD-3 criteria that undergo a successful 8 weeks acute medication stop, and does not overuse medication in the following 28 day period.
* Use of concurrent TTH preventive medication, with the exception of stable dose (≥3 months or 5 half-lives, whichever is longer) monotherapy of TTH preventive medication.
* Use of prophylactic medication with known prophylactic effect on other headache disorders, whatever the indication, with the exception of stable dose (≥3 months or 5 half-lives, whichever is longer) monotherapy of any preventive medication.
* Subjects taking opioids (>3 days per month) or barbiturates at the time of screening.
* Reduced sensibility, hearing or vision to a degree that impairs proper use of the app.
* Patients with comorbid psychiatric disorders with psychotic or other symptoms making compliance with the study protocol difficult, at the discretion of the investigator.
* Patients exhibiting a high degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator.
* Use of non-pharmacological preventive treatment, that in the opinion of the investigator is likely to interfere with the evaluation of the biofeedback treatment strategy under investigation. Stable non-pharmacological treatments for other indications than TTH that is not likely to interfere, is allowed if it is kept unaltered during study participation.
* Previous or current use of biofeedback equipment.
* Other pain conditions, not intended to be treated in this study, that in the opinion of the investigator could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints
* High probability neurological deterioration due to other medical conditions, that in the opinion of the investigator may confound outcome assessment.
* Have within 6 months of enrolment a significant untreated addiction to dependency-producing medications, alcohol, or illicit drugs.
* Abnormal pain behaviour, inappropriate medication-use and/or unresolved psychiatric illness, that in the opinion of the investigator are significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome.
* Subject is currently participating or planning to participate in another clinical investigation.
* Subject who is unlikely to follow Clinical Investigation Plan or where treatment seems futile in the opinion of the Investigator or have demonstrated an inability to sufficiently adhere to headache diary entries (<70%).

This study excludes patients with more than 1 migraine attack per month. A migraine attack is defined according to ICHD-3 criteria as attacks of unilateral, pulsating, moderate or severe headache lasting 4-72 hours that is aggravated by physical activity, associated with nausea and/or photophobia and phonophobia, and, in some cases, preceded by unilateral, fully-reversible central nervous system symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the efficacy of Cerebri-TTH in treatment group as compared to wait list control group in reducing the area under-the-headache curve (AUC) | From day 1 up to 38 weeks.
  Difference in the mean AUC from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group
To describe the treatment-emergent adverse events encountered during the investigation (include treatment emergent adverse events, ADEs, SADEs, and USADEs). | From randomization day-1 up to 34 weeks.
  A description of the frequency and severity of treatment- emergent adverse events, ADEs, SADEs, and USADEs).

SECONDARY OUTCOMES:
To investigate the efficacy of Cerebri-TTH in treatment group as compared to wait list control group in reducing the number of TTH days | From day 1 up to 38 weeks.
  Difference in number of days with TTH per 4 weeks in the baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group
To investigate the efficacy of Cerebri-TTH in treatment group as compared to wait list control group in reducing mean headache intensity | From day 1 up to 38 weeks.
  Difference in mean headache intensity from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group.
To investigate the efficacy of Cerebri-TTH in treatment group as compared to wait list control group in reducing mean headache duration. | From day 1 up to 38 weeks.
  Difference in mean headache duration from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group.
To investigate the efficacy of Cerebri-TTH in treatment group as compared to wait list control group in reducing the use of rescue medication | From day 1 up to 38 weeks.
  Difference in use of rescue medication from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group
To investigate patient-reported impact of headaches and headache treatment in the treatment group as compared to the control group. | From day 1 up to 38 weeks.
  Difference in mean HURT-3 score in the treatment group as compared to the wait-list control group.
To investigate patient-reported symptoms of anxiety and depression in the treatment group as compared to the control group. | From day 1 up to 38 weeks.
  Difference in mean Hospital Anxiety and Depression score (HADs) in the treatment group as compared to the wait-list control group.
To investigate the proportion of participants with at least 30% reduction in TTH duration and/or intensity from baseline to treatment between the treatment and control groups. | From day 1 up to 38 weeks.
  Difference in number of treatment responders (≥ 30% reduction in the mean AUC) from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group
To determine the frequency of device deficiencies | From randomization day 1 up to 34 weeks.
  Occurrence of device deficiencies.
Determine fetal outcome and the frequency of pregnancy complications | From day 1 up to 38 weeks.
  Occurrence of pregnancy complications and report fetal outcome data

OTHER OUTCOMES:
To investigate the proportion of participants with at least 50% reduction in TTH duration and/or intensity from baseline to treatment between the treatment and control groups. | From day 1 up to 38 weeks.
  Difference in number of treatment responders (≥ 50% reduction in the mean AUC)from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group.
To investigate the proportion of participants with at least 75% reduction in TTH duration and/or intensity from baseline to treatment between the treatment and control groups | From day 1 up to 38 weeks.
  Difference in number of treatment responders (≥ 75% reduction in the mean AUC) from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group.
To investigate the proportion of participants with at least 100% reduction in TTH duration and/or intensity from baseline to treatment between the treatment and control groups | From day 1 up to 38 weeks.
  Difference in number of treatment responders (100% reduction in the mean AUC) from baseline to the last 28-day period during the treatment phase, in the treatment group as compared to the wait-list control group.
Patient preference for treatment | From day 1 up to 38 weeks.
  12 weeks post-intervention the participant is asked to rate a benefit/tolerability ratio on an 11 point NRS scale. Similarly, a benefit/feasibility score will be assessed on a similar 11 point scale
To explore the effect of the treatment on patients self-reported sleep quality. | From day 1 up to 38 weeks.
  Difference in Bergen insomnia scale score (BIS) in the treatment group as compared to the wait-list control group. Participants state the number of days in which they experienced various sleep problems in the last month between 0 and 7 on an 8-point scale. The lowest score that can be taken from the scale is 0 and the highest score is 42.
To explore headache status in the 12 week extension period after completed 12 week biofeedback treatment | From day 1 up to 38 weeks.
  Development in headache endpoint variables in the 12 week eDiary extension period
To explore efficacy combining biofeedback arm and extension biofeedback arm data | From day 1 up to 38 weeks.
  Combined change in headache endpoint variables from baseline (last 28 period) before biofeedback treatment
To assess the subjective perception of treatment effectiveness from the patient's perspective. | From randomization day 1 up to 34 weeks
  Change in PGI-C at week 4, 8 and 12 in the intervention arm.
To assess the patient's self-perceived overall improvement in their condition after treatment | From randomization day 1 up to 34 weeks
  Change in PGI-I at week 4, 8 and 12 in the intervention arm.
To evaluate the level of perceived stress experienced by participants | From day 1 up to 38 weeks
  Mean change in PSS-14 total score from baseline to week12.

CONTACTS AND LOCATIONS:
Overall Officials: Tore Wergeland Meisingset, MD, PhD, Assc. Prof., Principal Investigator — Helse Nordtrøndelag Trust

IPD SHARING:
Plan to Share IPD: Undecided